CLINICAL TRIAL: NCT06357299
Title: Assessing Better Bottles for Babies (AB3)
Brief Title: Assessing Better Bottles for Babies
Acronym: AB3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Pro00115060
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-04

CONDITIONS: Pediatric Obesity; Weight Gain Trajectory; Infant Obesity
MeSH Terms: conditions — Pediatric Obesity; Body-Weight Trajectory

STUDY DESIGN:
Intervention Model Description: 2x2 factorial design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard, Clear (Experimental): This group will receive standard-sized clear bottles
  Interventions: Behavioral: Standard Bottle Size; Behavioral: Clear Bottle
- Standard, Opaque (Experimental): This group will receive standard-sized opaque bottles
  Interventions: Behavioral: Standard Bottle Size; Behavioral: Opaque Bottle
- Small, Clear (Experimental): This group will receive small-sized clear bottles
  Interventions: Behavioral: Small Bottle Size; Behavioral: Clear Bottle
- Small, Opaque (Experimental): This group will receive small-sized opaque bottles
  Interventions: Behavioral: Small Bottle Size; Behavioral: Opaque Bottle

INTERVENTIONS:
Behavioral: Small Bottle Size — Small sized bottle
  Arms: Small, Clear; Small, Opaque
Behavioral: Standard Bottle Size — Standard sized bottle
  Arms: Standard, Clear; Standard, Opaque
Behavioral: Clear Bottle — Clear bottle
  Arms: Small, Clear; Standard, Clear
Behavioral: Opaque Bottle — Opaque bottle
  Arms: Small, Opaque; Standard, Opaque

SUMMARY:
This study will use a 2 x 2 factorial design to test impact of two intervention strategies (bottle size and bottle opacity) on infant weight gain.

DETAILED DESCRIPTION:
Infants who gain weight rapidly have over 4 times higher odds of developing obesity as a child or adult; infants who are predominantly bottle-fed are at higher risk for excessive infancy weight gain and childhood obesity, yet there are not effective interventions to reduce excessive weight gain among infants who are bottle-fed. The investigators' preliminary work suggest that two novel intervention strategies are feasible and may reduce excessive infancy weight gain: reducing bottle size; and increasing bottle opacity. The investigators aim to test the independent and joint efficacy of these two intervention components among exclusively bottle-fed infants in a randomized, full factorial clinical trial. The investigators' primary objective is to measure the change in conditional weight gain z-score (CWGz) from birth to four months by study group. 4 groups are composed of two conditions: smaller bottles and opaque bottles, independently and in combination, via a 2x2 factorial trial design.

ELIGIBILITY:
Inclusion Criteria:

* Child is 3 days old to 1 month old
* Greater than 37 weeks gestational age at birth
* Birth weight greater than 3% for sex-specific WHO growth standard
* Caregiver must plan to use local clinic as infant's primary medical home for first 6 months of life
* Caregiver must speak English or Spanish as primary preferred language
* Caregiver age 18 years or older
* Caregiver must agree to use intervention bottles assigned during randomization and agree to stop using their existing bottles during the study period

Exclusion Criteria:

* Multiple gestation
* Significant congenital anomaly or acquired or inherited condition directly affecting feeding, physiology, metabolism, or growth
* Feeding with soy-based, hydrolyzed, lactose-reduced, or elemental formula
* Weight loss greater than 95% for population reference in the first two weeks of life

Ages: 3 Days to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Conditional weight gain z-score changes (CWGz) | Birth to 4 months
  CWGz scores will be calculated for each participant as the residual of the actual weight-for-age z-score at 4 months minus its predicted z-score from linear regression of the 4 month z-score on birth weight z-score. Intent-to-treat analyses will include regression models, stratified by sex, with CWGz score as the outcome.

SECONDARY OUTCOMES:
Formula volume per feed | Birth to 4 months
  At the time of in-home video recordings, the volume per feed will be measured from the pre- and post-weight of bottles by a food-grade scale calibrated and accurate to the nearest 0.01g.
Caregiver sensitivity to cues as measured by the Nursing Child Assessment Feeding Scale (NCAFS) | Birth to 4 months
  The Nursing Child Assessment Feeding Scale (NCAFS) measures discrete behaviors scored as "presence" or "absence" of each behavior/item. We will calculate feeding behavior scores on the "Sensitivity to Cues" subscale (score range 0 to 16) and "Responsiveness to Caregiver" subscale (score range 0 to 11). Score of 0 on a subscale means that none of the behaviors/items were observed, higher scores indicate more behaviors on the subscale were observed.

CONTACTS AND LOCATIONS:
Overall Officials: Charles T Wood, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No